CLINICAL TRIAL: NCT00400842
Title: A Double-blind, Placebo-controlled, Parallel-group, Comparative Study to Confirm the Safety and Efficacy of Oral 1.5 g/Day and 3.0 g/Day of SA-001 in Patients With Pancreatic Exocrine Insufficiency Caused by Chronic Pancreatitis or by Pancreatectomy
Brief Title: A Study of SA-001 to Treat Pancreatic Exocrine Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Toshiaki Yamaguchi, Sr. Clinical Program Manager, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S245.3.122
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Exocrine Pancreatic Insufficiency, Chronic Pancreatitis
Keywords: SA-001; Pancreatic Exocrine Insufficiency; Pancreatectomy
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- L (Experimental)
  Interventions: Drug: SA-001
- H (Experimental)
  Interventions: Drug: SA-001
- P (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SA-001 — 0.25 g of SA-001 pellets/capsule, 12 capsules/day for 7 days
  Arms: L
Drug: SA-001 — 0.25 g of SA-001 pellets/capsule, 6 capsules/day for 7 days
  Arms: H
Drug: Placebo — Placebo
  Arms: P

SUMMARY:
This study is to verify the efficacy of 3.0 g/day of SA-001 in patients with pancreatic exocrine insufficiency caused by chronic pancreatitis in the non-compensatory stage or by pancreatectomy as compared with placebo under a double-blind design using the change in a coefficient of fat absorption as a primary endpoint.

ELIGIBILITY:
Inclusion Criteria

* Subjects with chronic pancreatitis in the non-compensatory stage or pancreatectomy
* Subjects whose CFA is 80% or less
* Subjects who are able to be hospitalized

Exclusion Criteria

* Subjects who are judged to be difficult to have at least 40 g/day of fat intake during course of the study
* Subjects who have a known allergy to porcine protein and/or any component of digestive enzyme preparations
* Subjects who are in the acute phase of chronic pancreatitis
* Subjects with non-pancreatic malabsorption syndrome
* Subjects with acute pancreatitis or ileus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in CFA from baseline to the end of double-blind treatment | 7 days after baseline

SECONDARY OUTCOMES:
Stool fat excretion, stool weight, stool frequency, nutritional parameters | 7 days after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Toshiaki Yamaguchi, BS Pharm, Study Director — Abbott
Locations (98):
- Japan (98):
  - Site Reference ID/Investigator# 59845, Aichi
  - Site Reference ID/Investigator# 59933, Aichi
  - Site Reference ID/Investigator# 59928, Akita
  - Site Reference ID/Investigator# 59983, Amori
  - Site Reference ID/Investigator# 59984, Amori
  - Site Reference ID/Investigator# 59569, Ehime
  - Site Reference ID/Investigator# 59938, Ehime
  - Site Reference ID/Investigator# 59571, Fukuoka
  - Site Reference ID/Investigator# 59572, Fukuoka
  - Site Reference ID/Investigator# 59812, Fukuoka
  - Site Reference ID/Investigator# 59826, Fukuoka
  - Site Reference ID/Investigator# 59848, Fukuoka
  - Site Reference ID/Investigator# 59922, Fukuoka
  - Site Reference ID/Investigator# 59923, Fukuoka
  - Site Reference ID/Investigator# 59980, Fukuoka
  - Site Reference ID/Investigator# 59932, Fukushima
  - Site Reference ID/Investigator# 59935, Fukushima
  - Site Reference ID/Investigator# 59930, Higashiibaraki
  - Site Reference ID/Investigator# 59929, Hiroshima
  - Site Reference ID/Investigator# 59968, Hiroshima
  - Site Reference ID/Investigator# 59972, Hiroshima
  - Site Reference ID/Investigator# 59827, Hokkaido
  - Site Reference ID/Investigator# 59939, Hokkaido
  - Site Reference ID/Investigator# 59969, Hokkaido
  - Site Reference ID/Investigator# 59974, Hokkaido
  - Site Reference ID/Investigator# 59981, Hokkaido
  - Site Reference ID/Investigator# 59982, Hokkaido
  - Site Reference ID/Investigator# 59576, Hyōgo
  - Site Reference ID/Investigator# 59830, Hyōgo
  - Site Reference ID/Investigator# 59847, Hyōgo
  - Site Reference ID/Investigator# 59907, Hyōgo
  - Site Reference ID/Investigator# 59908, Hyōgo
  - Site Reference ID/Investigator# 59566, Ishikawa
  - Site Reference ID/Investigator# 59911, Ishikawa
  - Site Reference ID/Investigator# 59931, Kagoshima
  - Site Reference ID/Investigator# 59564, Kanagawa
  - Site Reference ID/Investigator# 59565, Kanagawa
  - Site Reference ID/Investigator# 59819, Kanagawa
  - Site Reference ID/Investigator# 59820, Kanagawa
  - Site Reference ID/Investigator# 59823, Kanagawa
  - Site Reference ID/Investigator# 59844, Kanagawa
  - Site Reference ID/Investigator# 59858, Kanagawa
  - Site Reference ID/Investigator# 59570, Kouchi
  - Site Reference ID/Investigator# 59574, Kumamoto
  - Site Reference ID/Investigator# 59854, Kurihara
  - Site Reference ID/Investigator# 59821, Kyoto
  - Site Reference ID/Investigator# 59910, Mie
  - Site Reference ID/Investigator# 59979, Mie
  - Site Reference ID/Investigator# 59849, Miyagi
  - Site Reference ID/Investigator# 59851, Miyagi
  - Site Reference ID/Investigator# 59857, Miyagi
  - Site Reference ID/Investigator# 59975, Miyagi
  - Site Reference ID/Investigator# 59976, Miyagi
  - Site Reference ID/Investigator# 59977, Miyagi
  - Site Reference ID/Investigator# 59937, Miyazaki
  - Site Reference ID/Investigator# 59913, Nagano
  - Site Reference ID/Investigator# 59825, Nagasaki
  - Site Reference ID/Investigator# 59814, Nagoya
  - Site Reference ID/Investigator# 59936, Nagoya
  - Site Reference ID/Investigator# 59927, Nara
  - Site Reference ID/Investigator# 59577, Okayama
  - Site Reference ID/Investigator# 59567, Osaka
  - Site Reference ID/Investigator# 59568, Osaka
  - Site Reference ID/Investigator# 59575, Osaka
  - Site Reference ID/Investigator# 59815, Osaka
  - Site Reference ID/Investigator# 59822, Osaka
  - Site Reference ID/Investigator# 59824, Osaka
  - Site Reference ID/Investigator# 59829, Osaka
  - Site Reference ID/Investigator# 59912, Osaka
  - Site Reference ID/Investigator# 59914, Osaka
  - Site Reference ID/Investigator# 59915, Osaka
  - Site Reference ID/Investigator# 59934, Osaka
  - Site Reference ID/Investigator# 59940, Osaka
  - Site Reference ID/Investigator# 59573, Saga
  - Site Reference ID/Investigator# 59556, Saitama
  - Site Reference ID/Investigator# 59925, Saitama
  - Site Reference ID/Investigator# 59555, Sapporo
  - Site Reference ID/Investigator# 59810, Shiga
  - Site Reference ID/Investigator# 59852, Shimane
  - Site Reference ID/Investigator# 59855, Suwa
  - Site Reference ID/Investigator# 59909, Tochigi
  - Site Reference ID/Investigator# 59557, Tokyo
  - Site Reference ID/Investigator# 59813, Tokyo
  - Site Reference ID/Investigator# 59818, Tokyo
  - Site Reference ID/Investigator# 59850, Tokyo
  - Site Reference ID/Investigator# 59859, Tokyo
  - Site Reference ID/Investigator# 59971, Tokyo
  - Site Reference ID/Investigator# 59973, Tokyo
  - Site Reference ID/Investigator# 59978, Tokyo
  - Site Reference ID/Investigator# 59816, Toyama
  - Site Reference ID/Investigator# 59970, Toyama
  - Site Reference ID/Investigator# 59811, Wakayama
  - Site Reference ID/Investigator# 59856, Yamagata
  - Site Reference ID/Investigator# 59926, Yamagata
  - Site Reference ID/Investigator# 59817, Yamaguchi
  - Site Reference ID/Investigator# 59924, Yamaguchi
  - Site Reference ID/Investigator# 59846, Yamanashi
  - Site Reference ID/Investigator# 59828, Yokohama